CLINICAL TRIAL: NCT00350025
Title: Randomized Phase II Trial of Cetuximab With and Without Weekly Paclitaxel in Patients With Previously Treated Advanced Urothelial Cancer
Brief Title: Study of Cetuximab With and Without Weekly Paclitaxel for Patients With Previously Treated Advanced Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-GU-004
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Urologic Neoplasm
Keywords: urothelial; urologic; neoplasm; advanced; metastatic
MeSH Terms: conditions — Urologic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab alone (Other): Cetuximab 250mg/m2 IV weekly during each 28 day cycle. Arm A closed to accrual June 11, 2009 for lack of efficacy
  Interventions: Drug: Cetuximab
- Cetuximab with Paclitaxel (Other): Paclitaxel 80 mg/m2 IV weekly for every 28 day cycle. Cetuximab 250mg/m2 IV weekly for every 28 day cycle.
  Interventions: Drug: Cetuximab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cetuximab — Cetuximab 250mg/m2 IV weekly for each 28 day cycle.
Drug: Paclitaxel — Paclitaxel 80mg/m2 IV weekly for each 28 day cycle.
  Other Names: Taxol
  Arms: Cetuximab with Paclitaxel

SUMMARY:
The purpose of this research study is to determine whether the investigational drug cetuximab, (Erbitux) alone or with paclitaxel (Taxol) can stabilize the growth of urothelial cancer.

DETAILED DESCRIPTION:
This research study is being done to find out if cetuximab, alone or with paclitaxel will slow the growth of urothelial cancers. Cetuximab is an antibody that blocks a protein called epidermal growth factor receptor (EGFR). EGFR sits on the outside of tumor cells and controls tumor cell growth. This agent has been looked at alone and with other chemotherapy drugs including paclitaxel. It has been found to be safe and can shrink other types of cancer.

This research study is also being done to find out if cetuximab, alone or with paclitaxel shrinks urothelial tumors. If it extends the time the tumors shrink. If it helps people live longer.

The purpose of this research study is to find out what effects (good and bad) these treatments have on you and your cancer. We do not know if you will benefit from this research study. It is possible that your condition will get better, but it is also possible that there will be no effect on your condition or that your condition will get worse. We can use what we learn from this research study to help other people with the same disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the urothelium (bladder,renal pelvis, ureter)
* Measurable disease by RECIST
* Patients who received only one prior systemic non-taxane regimen for urothelial cancer. May have received this in the adjuvant or neoadjuvant setting or for advanced disease.
* Signed IRB approved consent
* Must have tissue available for EGFR assessment and additional correlative studies
* ECOG PS 0-2
* 18 years of age or older
* Not of child bearing potential or negative pregnancy test within 7 days of treatment
* ANC greater than or equal to 1,500/ul
* Platelets greater than or equal to 100,00/ul
* Creatinine less than or equal to 2x institutional ULN or create. clearance greater than or equal to 30, bilirubin less than or equal to 1.5x ULN, AST&ALT less than or equal to 5x ULN

Exclusion Criteria:

* Received more than one prior regimen for advanced disease
* Prior radiation to more than 30% of marrow containing skeleton
* Prior therapy that specifically and directly targets the EGFR pathway
* Prior severe infusion reaction to a monoclonal antibody, pre-existing neuropathy greater than or equal to grade 2
* Prior reaction to Cremophor EL
* Known acute hepatitis B or C or known HIV
* Active or uncontrolled infection
* Significant history of uncontrolled cardiac disease
* Any concurrent chemotherapy not indicated in this study; or
* Any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ning Wong, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Wong YN, Litwin S, Vaughn D, Cohen S, Plimack ER, Lee J, Song W, Dabrow M, Brody M, Tuttle H, Hudes G. Phase II trial of cetuximab with or without paclitaxel in patients with advanced urothelial tract carcinoma. J Clin Oncol. 2012 Oct 1;30(28):3545-51. doi: 10.1200/JCO.2012.41.9572. Epub 2012 Aug 27. PMID 22927525

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Cetuximab Treatment Arm: Cetuximab 250mg/m2 IV weekly during each 28 day cycle. Arm A closed to accrual June 11, 2009 for lack of efficacy
  Cetuximab: Cetuximab 250mg/m2 IV weekly for each 28 day cycle.
- Arm B Paclitaxel and Cetuximab Combination Treatment Arm: Paclitaxel 80 mg/m2 IV weekly for every 28 day cycle. Cetuximab 250mg/m2 IV weekly for every 28 day cycle.
  Cetuximab: Cetuximab 250mg/m2 IV weekly for each 28 day cycle.
  Paclitaxel: Paclitaxel 80mg/m2 IV weekly for each 28 day cycle.
Period: Overall Study
Arm/Group | Arm A - Cetuximab Treatment Arm | Arm B Paclitaxel and Cetuximab Combination Treatment Arm
Started | 11 | 30
Completed | 11 | 28
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Cetuximab Treatment Arm | Arm B Paclitaxel and Cetuximab Combination Treatment Arm | Total
Number analyzed (Participants) | 11 | 28 | 39
Age, Continuous [Median (Full Range); unit: years] | 70 [49 to 83] | 69 [46 to 82] | 69 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 9 | 21 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 9 | 22 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Performance Status [Number; unit: participants] — ECOG scale of performance status was used to determine the ability of the patients to perform their daily functions.
  Grade(0)- Fully active Grade (1)- Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature Grade (2)- Ambulatory and capable of all selfcare but unable to carry out any work activities Grade (3)- Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours Grade (4) -Completely disabled Grade (5)- Dead
  participants
    0-1 | 11 | 25 | 36
    2 | 0 | 3 | 3
Primary site, No. of patients [Count of Participants; unit: Participants]
  Bladder | 9 | 26 | 35
  Renal Pelvis | 2 | 2 | 4
Previous Chemotherapy, No. of Patients [Count of Participants; unit: Participants]
  Gemcitabine and Platinum | 11 | 26 | 37
  MVAC | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Time Frame: Measures by CT scans following each 2 cycles of treatment and about every 8 weeks after off treatment for disease progression. Follow up for survival until time of death.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A - Cetuximab Treatment Arm | Arm B Paclitaxel and Cetuximab Combination Treatment Arm
Number analyzed (Participants) | 11 | 28
weeks | 7.6 [6 to NA] — The single agent cetuximab arm was closed for futility | 16.4 [12 to 25.1]

2. Secondary Outcome: Response Rate, Duration of Response, Time to Progression Will be Assessed With Radiographic Imaging
Time Frame: Measured by CT scans after every 2 cycles of treatment (about every 8 weeks)
Population: Overall Survival
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A - Cetuximab Treatment Arm | Arm B Paclitaxel and Cetuximab Combination Treatment Arm
Number analyzed (Participants) | 11 | 28
weeks
  Overall Survival | 17 [14.3 to NA] — The single-agent cetuximab arm was closed for futility | 42 [30.4 to 78]
  Overall Response Rate | NA [NA to NA] — The single-agent cetuximab arm was closed for futility | 25 [11 to 45]

ADVERSE EVENTS:
Arm/Group | Arm A - Cetuximab Treatment Arm | Arm B Paclitaxel and Cetuximab Combination Treatment Arm
Serious Adverse Events (participants affected / at risk) | 4/11 | 15/28
Other Adverse Events (participants affected / at risk) | 11/11 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Cetuximab Treatment Arm (N=11) | Arm B Paclitaxel and Cetuximab Combination Treatment Arm (N=28)
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Fever (Gastrointestinal disorders) | 1 | 0
death (General disorders) | 2 | 2
Urinary tract obstruction (Reproductive system and breast disorders) | 0 | 1
acute renal faliure (Renal and urinary disorders) | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 0 | 2
urinary retention (Renal and urinary disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
congestive heart faliure (Cardiac disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Infusion reaction (General disorders) | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1
hepatic faliure (Hepatobiliary disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 3
dehydration (Metabolism and nutrition disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
urosepsis (Injury, poisoning and procedural complications) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 3
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0
Rash (Immune system disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Cetuximab Treatment Arm (N=11) | Arm B Paclitaxel and Cetuximab Combination Treatment Arm (N=28)
Hemoglobin (Blood and lymphatic system disorders) | 10 | 25
ANC (Blood and lymphatic system disorders) | 1 | 12
Platelets (Blood and lymphatic system disorders) | 0 | 3
Leukocytes (Blood and lymphatic system disorders) | 3 | 20
Edema (Blood and lymphatic system disorders) | 2 | 12
DVT (Vascular disorders) | 0 | 2
Hypertension (Cardiac disorders) | 6 | 10
Dizziness (Nervous system disorders) | 0 | 8
fever (General disorders) | 2 | 5
fatigue (General disorders) | 8 | 27
chills (General disorders) | 2 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 16
Nail Loss (Skin and subcutaneous tissue disorders) | 0 | 4
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 10 | 27
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 10
Hemorrhage (Gastrointestinal disorders) | 1 | 11
vomiting (Gastrointestinal disorders) | 2 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 8 | 17
Diarrhea (Gastrointestinal disorders) | 3 | 12
Weight loss (Investigations) | 1 | 4
Ascites (Gastrointestinal disorders) | 0 | 1
confusion (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 11
Depression (Nervous system disorders) | 1 | 7
Neuropathy-motor (Nervous system disorders) | 1 | 3
Neuropathy - sensory (Nervous system disorders) | 4 | 11
Paresthesia (Nervous system disorders) | 4 | 10
Restlessness (Psychiatric disorders) | 1 | 0
Blurred vision (Eye disorders) | 0 | 2
Headache (General disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 10
cough (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 16
Alpkaline Phosphatase (Investigations) | 5 | 12
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4
hyperkalemia (Metabolism and nutrition disorders) | 3 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 17
blood bilirubin increase (Investigations) | 0 | 1
SGOT (Investigations) | 2 | 7
SGPT (Investigations) | 2 | 5
hepatic faliure (Hepatobiliary disorders) | 0 | 1
creatinine (Investigations) | 6 | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 23
Hematuria (Renal and urinary disorders) | 1 | 6
Infection (Infections and infestations) | 6 | 15
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 20
hypercalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 12
hyponatremia (Metabolism and nutrition disorders) | 0 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Mucositis (Gastrointestinal disorders) | 1 | 10
Dysgeucia (Nervous system disorders) | 1 | 8
Anorexia (Metabolism and nutrition disorders) | 5 | 14
Nausea (Gastrointestinal disorders) | 4 | 12
urinary retention (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes